CLINICAL TRIAL: NCT01695356
Title: A Double Blind Randomized Study Comparing the Ultraviolet (UV) Photoprotection With UV Plus Visible Light Photoprotection in the Treatment of Melasma.
Brief Title: Ultraviolet and UV-Visible Light Photoprotection for the Treatment of Melasma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidad Autonoma de San Luis Potosí (Other)
Collaborators: Hospital Central "Dr. Ignacio Morones Prieto" (Other)
Responsible Party: Principal Investigator, Juan Pablo Castanedo-Cazares, Dermatology assistant professor, Universidad Autonoma de San Luis Potosí
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VISUV-melasma
Record Dates: First submitted 2012-09-25; First posted 2012-09-28 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Melasma
Keywords: Melasma; sunscreens; visible light; ultraviolet light
MeSH Terms: conditions — Melanosis | interventions — Sunscreening Agents; octocrylene; titanium dioxide; Shade UVAGuard; bis-ethylhexyloxyphenol methoxyphenyl triazine; drometrizole trisiloxane; octyl triazone; terephthalylidene dicamphor sulfonic acid; oxybenzone; octylmethoxycinnamate; Zinc Oxide; ferric oxide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 290-400 nm sunscreen (Active Comparator): Sunscreen containing Mexoryl SX, Mexoryl XL, Titanium Dioxide, Octocrylene, Tinosorb S, Avobenzone, and Ethylhexyl triazone.
  Fluid vehicle administered daily, from 8AM to 5PM every 3 hr, for 12 weeks.
  Interventions: Drug: 290-400 nm sunscreen
- 290-800 nm sunscreen (Experimental): Sunscreen containing Benzophenone-3, Octinoxate, Octocrylene, Titanium Dioxide, Zinc Oxide, and iron oxide.
  Fluid vehicle administered daily, from 8AM to 5PM every 3 hr, for 12 weeks.
  Interventions: Drug: 290-800 nm sunscreen

INTERVENTIONS:
Drug: 290-400 nm sunscreen — A broad UV spectrum sunscreen will be applied every 3 hours for 12 weeks. The affected surface will be covered with a 2 mg/cm^2 layer of the product as indicated on the affected areas of the face.
  Other Names: Octocrylene; Titanium dioxide; Butyl methoxydibenzoylmethane; Bis-ethylhexyloxyphenol methoxyphenyl triazine; Drometrizole trisiloxane; Ethylhexyl triazone; Terephthalylidene dicamphor sulfonic acid
  Arms: 290-400 nm sunscreen
Drug: 290-800 nm sunscreen — A UV-visible light spectrum sunscreen will be applied every 3 hours for 12 weeks. The affected surface will be covered with a 2 mg/cm^2 layer of the product as indicated on the affected areas of the face.
  Other Names: Benzophenone-3; Octinoxate; Octocrylene; Titanium Dioxide; Zinc Oxide; Iron oxide
  Arms: 290-800 nm sunscreen

SUMMARY:
Melasma is an acquired discoloration of the skin characterized by brown colour changes commonly on the face. The duration of this double-blind clinical trial will be 12 weeks. The control group will receive treatment with topical Hydroquinone (4%) and a Broad spectrum UV sunscreen. The experimental group, 4% topical hydroquinone and a Broad spectrum UV-visible light sunscreen. Visible light has melanotic properties and avoiding it can be part of the treatment for melasma patients. The estimated number of subjects to be recruited and randomized for the study is at least 25 per group. The purpose of this study is determine if there is a difference in the improvement between these two sunscreens types. Melasma Area and Severity Index (MASI) score will be assessed at the beginning of the study and at weeks 4, 8, and 12. Photographs, colorimetry and histological assessment will be also evaluated. Occurrence of adverse effects will also be recorded.

DETAILED DESCRIPTION:
Melasma is a common acquired hypermelanosis in dark skin populations, usually characterized by symmetrical, irregular macules occurring in photo-exposed areas such as face. Treatment with sunscreens and depigmenting compounds such as hydroquinone, are still the gold standard in this condition.

Visible light has pigmenting properties that could be interfering with the treatment in melasma patients. So, the primary objective of this study is to compare the depigmenting adjuvant effect of using a UV-visible blocking sunscreen against a UV sunscreen.

Patients who are included in the study will be randomly assigned to receive one of the sunscreen type, which should use for 12 weeks. The sun blocking agents should be applied in the affected regions every 3 hours from 8AM to 5PM. The evaluation of clinical improvement will be done in a blinded modality by means of the MASI score, the Global Physician Assessment, as well as colorimetry and histological melanin content. Evaluations will be held on visits at 4, 8 and 12 weeks. Skin biopsy will be taken at onset and at 12 weeks.

At the end of the study, data will be compared concerning the former parameters. All side effects will be recorded and analysed.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Women over 25 years of age
* Dermatologic diagnostic of melasma
* Phototype III or more

Exclusion Criteria:

* Pregnant or breastfeeding
* Postbirth, abortion in the past 6 months
* Having an endocrine or autoimmune disease
* Under hormonal therapy of any kind including contraceptives or it´s use in the past 6 months
* Currently under treatment for melasma including sunscreens
* Currently under radiation therapy, chemotherapy, immunosuppressants of any kind or phototherapy or it´s use in the past 6 months
* Having used or are consuming photosensitizing substances, oral or topical

Ages: 25 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2012-09; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Depigmentation of melasma lesions by Colorimetry | 12 weeks
  Quantification of the colour change in the melasma lesions by means of the L axis of the CIE system. 0 value is pure white, 100 value is total black.

SECONDARY OUTCOMES:
MASI (Melasma Area Severity Index) | 12 weeks
  It is a clinical instrument of melasma measurement. The total score would range from 0-24, involving the forehead (30%), right malar (30%), left malar (30%) and chin (10%), and using area of involvement (0=absent, 1=<10%, 2=10%-29%, 3=30%-49%, 4=50%-69%, 5=70%-89% and 6=90%-100%) and darkness (0=absent, 1=slight, 2=mild, 3=marked and 4=severe). Computation would be as follows: 0.3 A(f) D(f) + 0.3 A(lm) D(lm) + 0.3 A(rm) D(rm) + 0.1 A(c) D(c).
Melanin content by histologic quantification. | 12 weeks
  The Fontana-Masson Stain is specific for melanin, this histochemical reaction reveals accumulations of black material wherever melanin is located. A skin biopsy of lesions will be taken initially and at the end of study. The melanin content will be quantified by a software image analysis of the slides.
Global Physician Assessment | 12 weeks
  Clinical improvement is assessed by means of digital photographic registration (frontal, right, and left views). An independent observer clinically graded the global improvement as poor (0-25%), mild (26-50%), good (51-75%), and excellent (>75%).

CONTACTS AND LOCATIONS:
Overall Officials: Diana Hernandez-Blanco, MD, Principal Investigator — Hospital Central "Dr. Ignacio Morones Prieto"; Juan P Castanedo-Cazares, MD, Study Director — Hospital Central "Dr. Ignacio Morones Prieto"; Bertha Torres-Alvarez, MD, Study Chair — Hospital Central "Dr. Ignacio Morones Prieto"
Locations (1):
- Dermatology Department. Hospital Central "Dr. Ignacio Morones Prieto", San Luis Potosí City, San Luis Potosí, Mexico

REFERENCES:
- [Background] Navarrete-Solis J, Castanedo-Cazares JP, Torres-Alvarez B, Oros-Ovalle C, Fuentes-Ahumada C, Gonzalez FJ, Martinez-Ramirez JD, Moncada B. A Double-Blind, Randomized Clinical Trial of Niacinamide 4% versus Hydroquinone 4% in the Treatment of Melasma. Dermatol Res Pract. 2011;2011:379173. doi: 10.1155/2011/379173. Epub 2011 Jul 21. PMID 21822427
- [Background] Torres-Alvarez B, Mesa-Garza IG, Castanedo-Cazares JP, Fuentes-Ahumada C, Oros-Ovalle C, Navarrete-Solis J, Moncada B. Histochemical and immunohistochemical study in melasma: evidence of damage in the basal membrane. Am J Dermatopathol. 2011 May;33(3):291-5. doi: 10.1097/DAD.0b013e3181ef2d45. PMID 21317614
- [Background] Moncada B, Sahagun-Sanchez LK, Torres-Alvarez B, Castanedo-Cazares JP, Martinez-Ramirez JD, Gonzalez FJ. Molecular structure and concentration of melanin in the stratum corneum of patients with melasma. Photodermatol Photoimmunol Photomed. 2009 Jun;25(3):159-60. doi: 10.1111/j.1600-0781.2009.00425.x. PMID 19438997
- [Background] Hernandez-Barrera R, Torres-Alvarez B, Castanedo-Cazares JP, Oros-Ovalle C, Moncada B. Solar elastosis and presence of mast cells as key features in the pathogenesis of melasma. Clin Exp Dermatol. 2008 May;33(3):305-8. doi: 10.1111/j.1365-2230.2008.02724.x. PMID 18419607
- [Background] Espinal-Perez LE, Moncada B, Castanedo-Cazares JP. A double-blind randomized trial of 5% ascorbic acid vs. 4% hydroquinone in melasma. Int J Dermatol. 2004 Aug;43(8):604-7. doi: 10.1111/j.1365-4632.2004.02134.x. PMID 15304189